CLINICAL TRIAL: NCT02657382
Title: Effects of Biofeedback on Myocardial Blood Flow Changes During Mental Stress in Patients With Coronary Artery Disease
Brief Title: Mental Stress Ischemia: Biofeedback Study
Acronym: MIBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB00083616
Record Dates: First submitted 2016-01-13; First posted 2016-01-15 (Estimated); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Cardiovascular Disease; Coronary Artery Disease
Keywords: Biofeedback; Myocardial Imaging
MeSH Terms: conditions — Cardiovascular Diseases; Coronary Artery Disease | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Heart Rate Variability (HRV) Biofeedback (BF) (Experimental): Participants with coronary artery disease randomized to this group will complete myocardial blood flow (MBF) imaging and mental stress tests. Participants in this group will also participate in heart rate variability (HRV) biofeedback (BF) during the first six weeks of the study.
  Interventions: Behavioral: Heart Rate Variability (HRV) Biofeedback (BF); Other: Mental Stress Protocol
- Waitlist Control (Experimental): Participants with coronary artery disease randomized to this group will complete myocardial blood flow (MBF) imaging and mental stress tests.Participants in this group will receive the heart rate variability (HRV) biofeedback (BF) intervention between the week 6 and week 12 study visits.
  Interventions: Behavioral: Heart Rate Variability (HRV) Biofeedback (BF); Other: Mental Stress Protocol

INTERVENTIONS:
Behavioral: Heart Rate Variability (HRV) Biofeedback (BF) — Heart Rate Variability (HRV) biofeedback involves deep breathing, mindfulness (focusing on one's emotions and thoughts) and cognitive therapy (identifying and changing unhelpful or inaccurate thinking and distressing emotional responses). It is a 6-week training with one hour sessions with a certified biofeedback coach once per week. A handheld personal stress reliever device will be provided to the patients to practice at home for 20 minutes a day.
Other: Mental Stress Protocol — Mental stress will consist of a 3-min math serial subtraction paradigm.The participants will be asked to serially subtract 7 from number specified by the researcher. For participants who have difficulty with this task, easier serial subtraction will be provided for. Throughout the task, to increase stressfulness and titrate difficulty, the participant will be prompted for faster performance and the starting number from which they were subtracting will be periodically changed. Finally, to add an evaluation component, participants will be given negative feedback during the test.

SUMMARY:
The purpose of this study is to evaluate the blood flow to the heart during stress and assess changes in blood flow after psychological treatment in participants with coronary artery disease. The aims of the study are to assess the effects of heart rate variability (HRV) biofeedback (versus usual care) on global and regional myocardial blood flow (MBF), peripheral vascular function, and autonomic changes during mental stress.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the blood flow to the heart during stress and assess changes in blood flow after psychological treatment in participants with coronary artery disease. This is a randomized controlled study. The aims of the study are to assess the effects of heart rate variability (HRV) biofeedback (versus usual care) on global and regional myocardial blood flow (MBF), peripheral vascular function, and autonomic changes during mental stress.

All participants will undergo myocardial flow/perfusion imaging with positron emission tomography (PET) imaging at rest and after a standardized arithmetic mental stress test. Participants will then undergo repeat testing after 6 weeks. At 12 weeks, participants will also undergo a limited examination without myocardial perfusion imaging. The intervention group will receive biofeedback after enrollment, and the wait-list control group will receive the intervention between week 6 and week 12 study visits (without imaging).

ELIGIBILITY:
Inclusion Criteria:

Prior participation in the Mental Stress Ischemia: Mechanisms and Prognosis (MIPS) study

Eligibility for the MIPS study included:

* Angiographically proven disease including at least 1 major vessel with evidence of disease but with no specific minimum lumen diameter criteria
* Prior myocardial ischemia (MI) (>1 months) documented by typical elevation of enzymes and typical pain or ECG changes
* Abnormal coronary intravascular ultrasound exam (IVUS) demonstrating atherosclerosis of at least 1 vessel
* Post bypass surgery or post PCI (percutaneous intervention)* (> 1 year after complete revascularization)
* Positive nuclear scan or stress exercise test

Exclusion Criteria:

* Unstable angina, myocardial infarction, decompensated congestive heart failure in past week
* Severe concomitant medical problems expected to shorten life expectancy to less than 5 years
* Pregnancy. Women of childbearing age who are not postmenopausal will be screened by pregnancy test
* Systolic blood pressure >190 mm Hg or diastolic blood pressure >115 mm Hg on the day of the test
* History of current alcohol or substance abuse or dependence (past year); or history of severe psychiatric disorder other than major depression, such as schizophrenia or psychotic depression
* For patients who are unable to exercise, we will do a pharmacological stress test with regadenoson. Additional exclusion criteria for regadenoson administration include second- or third-degree AV block (without permanent pacemakers) and bronchospastic disease such as asthma or severe chronic obstructive lung disease
* Weight more than 450 lbs or a body habitus that is unfit for the nuclear camera dimensions
* Inflammatory diseases - Rheumatoid Arthritis, Lupus, Hepatitis, HIV, Crohn's, etc.
* Dialysis
* Any malignancy (No active/any metastasis from oncology notes)
* Dementia/Alzheimer's
* Drug incompliance
* No supporting documents for CAD history
* Permanent atrial fibrillation
* Clean vessels after revascularization
* Any transplants
* On any immunosuppressants
* Immobile, in wheel chair (If patient can lift self out of wheel chair then it is okay)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2020-06-24 (Actual); Study Completion 2020-06-24 (Actual)

PRIMARY OUTCOMES:
Change in Global Myocardial Perfusion During Mental Stress | Baseline, Week 6
  Global myocardial perfusion during mental stress will be tested via positron emission topography (PET) scan while completing the mental stress protocol.
Change in Regional Myocardial Perfusion During Mental Stress | Baseline, Week 6
  Regional myocardial perfusion during mental stress will be tested via positron emission topography (PET) scan while completing the mental stress protocol.

SECONDARY OUTCOMES:
Change in Arterial Compliance assessed by Augmentation Index and Pulse Wave Velocity | Baseline, Week 12
  Arterial compliance will be assessed using the SphygmaCor device which is a non-invasive method for assessing the cardiovascular system focused on central blood pressures, measures of arterial stiffness and autonomic function. Peripheral pressure waveforms are recorded from the radial artery at the wrist, using applanation tonometry with a high-fidelity micromanometer. After 20 sequential waveforms have been acquired, a validated generalized transfer function will be used to generate the corresponding central aortic pressure waveform.
Change in Number of Ischemic Regions | Baseline, Week 6
  Number of ischemic regions will be measured by PET scan myocardial infusion. Change is defined as the difference in the number of ischemic regions from baseline compared to week six.
Change in Peripheral Arterial Tonometry (PAT) Ratio | Baseline, Week 12
  The Peripheral Arterial Tonometry (PAT) reflects the magnitude of change in finger-tip blood flow induced by mental stress by measuring the ratio of pulse wave amplitude during mental stress compared to rest.
Change in Resting Norepinephrine Levels | Baseline, Post Intervention (Up to 12 weeks)
  Change in resting norepinephrine levels post mental stress test will be evaluated via blood draws obtained at baseline, immediately post mental stress testing, and 90 minutes post mental stress testing. Testing will be completed at all study visits. Change is measured as the difference between resting norepinephrine levels at baseline and post intervention.
Change in Resting Epinephrine Levels | Baseline, Post Intervention (Up to 12 weeks)
  Change in resting epinephrine levels post mental stress test will be evaluated via blood draws obtained at baseline, immediately post mental stress testing, and 90 minutes post mental stress testing. Testing will be completed at all study visits. Change is measured as the difference between resting epinephrine levels at baseline and post intervention.
Change in Resting Dopamine Levels | Baseline, Post Intervention (Up to 12 weeks)
  Change in resting dopamine levels post mental stress test will be evaluated via blood draws obtained at baseline, immediately post mental stress testing, and 90 minutes post mental stress testing. Testing will be completed at all study visits. Change is measured as the difference between resting dopamine levels at baseline and post intervention.
Change in Flow-Mediated Dilation (FMD) of the Brachial Artery | Baseline, Week 12
  Two-dimensional ultrasound images will be used to assess flow-mediated dilation (FMD) of the brachial artery before and 30 minutes after mental stress testing. Images will be obtained with an Acuson 10 mHz linear array transducer and an Acuson Aspen ultrasound system. Change is measured as the difference in FMD at baseline and week 12.

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Emory University Hospital, Atlanta, Georgia
  - Emory University, Atlanta, Georgia
  - Rollins School of Public Health, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia

REFERENCES:
- [Derived] Shah AJ, Raggi P, She H, Quyyumi AA, Levantsevych O, Johnson M, Schmidt K, Garcia E, Piccinelli M, Abdulbaki R, Abdelhadi N, Kaseer B, Ginsberg JP, Vaccarino V, Bremner JD. Heart Rate Variability Biofeedback and Mental Stress Myocardial Flow Reserve: A Randomized Clinical Trial. JAMA Netw Open. 2025 Oct 1;8(10):e2538416. doi: 10.1001/jamanetworkopen.2025.38416. PMID 41118163
- [Derived] Gurel NZ, Carek AM, Inan OT, Levantsevych O, Abdelhadi N, Hammadah M, O'Neal WT, Kelli H, Wilmot K, Ward L, Rhodes S, Pearce BD, Mehta PK, Kutner M, Garcia E, Quyyumi A, Vaccarino V, Raggi P, Bremner JD, Shah AJ. Comparison of autonomic stress reactivity in young healthy versus aging subjects with heart disease. PLoS One. 2019 May 8;14(5):e0216278. doi: 10.1371/journal.pone.0216278. eCollection 2019. PMID 31067240